CLINICAL TRIAL: NCT02577328
Title: Pain Management in Internal Medicine Department
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Bnai Zion Medical Center (Other Government)
Responsible Party: Principal Investigator, Maayan.Ben Sasson, Dr., Bnai Zion Medical Center
Other Study IDs: 0138-14-BNZ
Record Dates: First submitted 2015-10-07; First posted 2015-10-16 (Estimated); Last update posted 2015-10-16 (Estimated); Status verified 2015-06

CONDITIONS: Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The assessment of pain management in Internal medicine department.

DETAILED DESCRIPTION:
The experimental procedure - A Literature review of the management of pain in internal departmnet and after that defining and identifying gaps between the pain management practice recommendations in the literatureareas to that of the departmnet.

Determining the educational processes for the medical team, in initiation treatment for pain and pain assessment. As well, obtain quality indicators to monitor pain management.

Assessment of attitudes, knowledge and tools for pain management team before the educational process and afterwards.

In patients with mild pain or above, a combination of quantitative and qualitative tools will assess the pain and its treatment along the hospitalization in the Internal medicine ward.

ELIGIBILITY:
Inclusion Criteria:

* All patient with mild pain and above

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All patients in the ward with mild pain and above
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2015-11; Primary Completion 2015-12 (Estimated); Study Completion 2016-07 (Estimated)

PRIMARY OUTCOMES:
pain reduction | during hospitalization (days)-up to7 days
  Reviewing the pain scale (VAS or other) of a patient with mild pain during the hospitalization